CLINICAL TRIAL: NCT04102358
Title: The Need for Supplemental Blocks in Single Versus Triple Injections in Infraclavicular Brachial Plexus Blocks With Medial Approach: A Clinical and an Anatomical Study
Brief Title: The Need for Supplemental Blocks in Infraclavicular Brachial Plexus Blocks
Status: Completed | Type: Observational
Sponsor: Derince Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Hande Gurbuz, Principal Investigator, Derince Training and Research Hospital
Other Study IDs: U1111-1240-8832
Record Dates: First submitted 2019-09-23; First posted 2019-09-25 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Anesthesia, Regional
Keywords: Vertical infraclavicular block; brachial plexus anatomy
MeSH Terms: interventions — Injections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Single injection: Patients who received an infraclavicular block with a single injection technique were included in Group-S.
  Interventions: Procedure: Medial approach infraclavicular block with single injection
- Triple injection: Patients who received an infraclavicular block with a triple injection technique were included in Group-T.
  Interventions: Procedure: Medial approach infraclavicular block with triple injection

INTERVENTIONS:
Procedure: Medial approach infraclavicular block with single injection — infraclavicular blocks performed with single injection
  Groups: Single injection
Procedure: Medial approach infraclavicular block with triple injection — infraclavicular blocks performed with triple injection
  Groups: Triple injection

SUMMARY:
Theoretically, all surgeries below mid-humerus can be done under infraclavicular (IC) blocks. Following the introduction of ultrasonography (USG) to clinical anesthesia, plexus, and nerve blocks under the guidance of USG have gained wide acceptance for the high rates of block success and low risk of complications (1). In this study, the main aim is to evaluate the single injection and triple injection techniques in IC blocks with a USG-guided medial approach in terms of block success and the need for supplementary blocks. The secondary goals are to compare the complication rates and sensory block durations and to discuss the possible reasons for the failure of the blocks.

DETAILED DESCRIPTION:
Theoretically all surgeries below mid-humerus can be done under infraclavicular (IC) blocks. Following the introduction of ultrasonography (USG) to the clinical anesthesia, plexus and nerve blocks under the guidance of USG have gained wide acceptance for the high rates of block success, and low risk of complications. At the same time, it was also shown that USG-guided IC blocks can shorten procedural times and accelerate the onset of the blocks.

Several methods for IC blocks have been described. Based on the anatomical knowledge, we hypothesized that in medial approaches the need for supplementary blocks would be low with single injections as well as triple injections. In this study, the main aim is to evaluate the single injection and triple injection techniques in IC blocks with a USG-guided medial approach in terms of block success and the need for supplementary blocks. The secondary goals are to compare the complication rates and sensory block durations and to discuss the possible reasons for the failure of the blocks.

Medical records of 139 patients scheduled for elective or emergent hand, wrist, forearm, elbow, and distal arm surgery were analyzed. Patients older than 14 years with ASA physical status I-III who underwent surgery between October 2017 and March 2019 were retrospectively evaluated. Exclusion criteria included non-cooperative patients, refusal of the regional anesthesia, known neuropathy that could prevent the evaluation of the efficacy of the block, different techniques used for infraclavicular brachial plexus blocks (lateral sagittal, coracoid, …etc.), and known allergy to local anesthetic drugs.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-III
* upper extremity surgery
* blocks were performed by the same anesthesiologist

Exclusion Criteria:

* non-cooperative patients
* refusal of the regional anesthesia
* known neuropathy
* different technique used for infraclavicular brachial plexus blocks (lateral sagittal, coracoid, …etc.)
* known allergy to local anesthetic drugs.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients underwent surgery for upper extremity under medial approach infraclavicular block between October 2017 and March 2019
Sampling Method: Non-Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Supplemented blocks | 1 hour
  30 minutes after the block, if one or two of the median, radial, ulnar or musculocutaneous nerves were still unblocked, these nerves were located either with a peripheric nerve stimulator or an ultrasound, in the axilla or on the more distal parts of their traces on arm and forearm and then supplemented.

SECONDARY OUTCOMES:
Complete Failure | 30 minutes
  If more than two of these nerves (median, radial, ulnar or musculocutaneous) were remained unblocked, no supplementary blocks were applied, then it was considered as having a failed block and general anesthesia was administered.
Recovery of sensory block | 24 hours
  the first time of the need for analgesics
Discomfort during IC block | 1 hour
  paresthesia during the infraclavicular block
Inadvertent vascular puncture | 1 hour
  inadvertent vascular puncture during the infraclavicular block

CONTACTS AND LOCATIONS:
Overall Officials: Tuncay Colak, Prof, Study Chair — Kocaeli University
Locations (1):
- Derince Training and Research Hospital, Kocaeli, Derince, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available within 6 months of study completion.
Access Criteria: Data access requests will be reviewed by the researchers. Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Background] Abrahams MS, Aziz MF, Fu RF, Horn JL. Ultrasound guidance compared with electrical neurostimulation for peripheral nerve block: a systematic review and meta-analysis of randomized controlled trials. Br J Anaesth. 2009 Mar;102(3):408-17. doi: 10.1093/bja/aen384. Epub 2009 Jan 26. PMID 19174373
- [Background] Li JW, Songthamwat B, Samy W, Sala-Blanch X, Karmakar MK. Ultrasound-Guided Costoclavicular Brachial Plexus Block: Sonoanatomy, Technique, and Block Dynamics. Reg Anesth Pain Med. 2017 Mar/Apr;42(2):233-240. doi: 10.1097/AAP.0000000000000566. PMID 28157792
- [Background] Kilka HG, Geiger P, Mehrkens HH. [Infraclavicular vertical brachial plexus blockade. A new method for anesthesia of the upper extremity. An anatomical and clinical study]. Anaesthesist. 1995 May;44(5):339-44. doi: 10.1007/s001010050162. German. PMID 7611581